CLINICAL TRIAL: NCT04900285
Title: Pilot Study for Feasibility of Using an Oral Appliance for Decreasing Snoring
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Norton Healthcare (Other)
Collaborators: Delta Dental Foundation (Other)
Responsible Party: Principal Investigator, David Winslow, Jr., MD, FCCP, Pulmonologist, Staff Physician, Norton Healthcare
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20-N0387
Record Dates: First submitted 2021-05-13; First posted 2021-05-25 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Snoring
MeSH Terms: conditions — Snoring

STUDY DESIGN:
Intervention Model Description: Subject serve as their own control sleeping without the device for five days and recording snoring on the SnoreLab app and filling out the Snore Outcomes Survey. The lower dental device is used for five days while recording snoring. The subject will then complete the Comfort and Difficulties Form and the bed partner completes the Snore Outcomes Survey. The process is repeated with the upper device for those who tolerate the lower device. use.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Dental Device Arm (Other): Subjects in this single arm study serve as their own control by recording snoring on the SnoreLab device for five days and completing the Snore Outcomes survey. After five nights with now device, the lower dental device is used for five nights and snoring is recorded in the SnoreLab app. At the end of the five nights the subjects complete the Comfort and Difficulties Form and the bed partner completes the Snore Outcomes Survey. If the lower device was tolerated well, the process is repeated with the upper dental device used with the lower device.
  Interventions: Device: Delta Dental Oral Device

INTERVENTIONS:
Device: Delta Dental Oral Device — The oral device is designed to move the genioglossus forward, with interior attachments to maintain the placement of the tongue on the floor of the mouth forward. In addition, bite plates made of the Ethylene-vinyl acetate (EVA) plastic were fabricated and embedded with the mouthpiece to encourage subjects to bite down and push the tongue under the interior lower attachment. The upper plate is made of the same material and slightly opens the bite to improve oral air flow further. The primary component of the mouthpiece is fabricated with Vistamaxx material, which is semi-crystalline 2mm co-polymer that can be molded by the user with Nurse assistance to provide a custom fit.
  The subject will be fitted by moistening and heating in a microwave. Tthe research staff member will assist to ensure proper fit with both the lower and upper dental devices.
  The subject then completes the data collection portion regarding using the SnoreLab app and survey completion as previously described.

SUMMARY:
This research study proposes to determine how well tolerated and effective lower and upper oral dental devices are at reducing snoring. The device is designed to move the genioglossus muscle forward, with interior attachment to maintain forward placement of of he tongue on the bottom of the mouth.

DETAILED DESCRIPTION:
This study proposed to determine if the use of an oral device which causes forward positioning of the tongue will decrease the intensity and frequency of snoring as measured by the SnoreLab phone app, evaluate the level of snoring as measured by the bed partner, evaluate tolerance and comfort of the device and evaluate the quality of sleep of the subject by the bed partner.

Subjects will sleep at home using the SnoreLab app to record snoring for five nights and fill out the Snore Outcomes Survey. They will then utilize the lower dental device for five nights recording their snoring. At the end of the five nights of using the lower dental device, the subjects will fill out the comfort and difficulties form with the bed partner completing the Snore Outcomes Survey. If the lower device is tolerated, the process is repeated with the upper device added to the lower device.

ELIGIBILITY:
Inclusion Criteria:

1. . Able to provide informed consent
2. Age 18 or older
3. Self-report of snoring problems
4. Has a bed partner that is willing and able to consent as well as answer questions related to partner's snoring both with and without oral device-

Exclusion Criteria:

1. Missing teeth.
2. Respiratory disorders requiring treatment including asthma, COPD
3. Poor dental health including gum disease or loose teeth
4. Dental implants placed within the last three months
5. Temporomandibular joint dysfunction
6. Presence of mouth or jaw pain
7. Bruxism (teeth grinding)
8. Full dentures
9. No bed partner
10. Braces
11. Diagnosed with Obstructive or Central Sleep Apnea, Sleep Apnea
12. Uncontrolled RLS
13. Ongoing or prior use of a dental device
14. Noise in bedroom i.e., fan, bed partner snoring
15. Other medical or sleep issues which will interfere with the device per PI discretion
16. Does not have a smart phone
17. Other medical condition that PI believes will make the patient ineligible for participation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Intensity of Snoring (Snore Lab App; range from Quiet to Epic snoring, Epic is a worse outcome) | Daily up to 15 days
  To determine if use of a device to position the tongue forward will decrease the intensity of snoring.
Frequency of Snoring (Snore Lab App, app records snoring through the night) | Daily up to 15 days
  To determine if use of a device to position the tongue forward will decrease the frequency of snoring.

SECONDARY OUTCOMES:
Partner Assessment of Snoring (Snore Outcomes Survey, response scale varies per item) | Day 5 (end of no device use)
  Evaluate the level of snoring of the subject by bed partner using approved questionnaire
Partner Assessment of Snoring (Snore Outcomes Survey, response scale varies per item) | Day 10 (end of lower device use)
  Evaluate the level of snoring of the subject by bed partner using approved questionnaire
Partner Assessment of Snoring (Snore Outcomes Survey, response scale varies per item) | Day 15 (end of lower and upper device use)
  Evaluate the level of snoring of the subject by bed partner using approved questionnaire
Device Tolerance and Comfort (Tolerance Form) | Day 5 (end of no device use)
  Subject Evaluation of tolerance and comfort of the oral device by questionnaire
Device Tolerance and Comfort (Tolerance Form) | Day 10 (end of lower device use)
  Subject Evaluation of tolerance and comfort of the oral device by questionnaire
Device Tolerance and Comfort (Tolerance Form) | Day 15 (end of lower and upper device use)
  Subject Evaluation of tolerance and comfort of the oral device by questionnaire
Quality of Sleep Assessment (Snore Outcomes Survey, response scale varies per item) ) | Day 5 (end of no device use)
  Evaluate the quality of sleep of subject by bed partner by questionnaire
Quality of Sleep Assessment (Snore Outcomes Survey, response scale varies per item) | Day 10 (end of lower device use)
  Evaluate the quality of sleep of subject by bed partner by questionnaire
Quality of Sleep Assessment (Snore Outcomes Survey, response scale varies per item) | Day 15 (end of lower and upper device use)
  Evaluate the quality of sleep of subject by bed partner by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: David Winslow, MD, Principal Investigator — Norton Healthcare
Locations (1):
- Norton Clinical Research Group, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No
No, this is a limited feasibility study and data will not be generalizable to the public due to small sample size. (n=30)

REFERENCES:
- [Background] American Academy of Sleep Medicine. International Classification of Sleep Disorders. 3rd ed. Darien, IL: American Academy of Sleep Medicine; 2014.
- [Background] Gliklich RE, Wang PC. Validation of the snore outcomes survey for patients with sleep-disordered breathing. Arch Otolaryngol Head Neck Surg. 2002 Jul;128(7):819-24. doi: 10.1001/archotol.128.7.819. PMID 12117343
- [Background] Meira e Cruz M., Cardiovascular Center of University of Lisbon, Lisbon School of Medicine, Lisbon, Portugal; Email: mcruz@medicina.ulisboa.pt
- [Result] Cooke ME, Battagel JM. A thermoplastic mandibular advancement device for the management of non-apnoeic snoring: a randomized controlled trial. Eur J Orthod. 2006 Aug;28(4):327-38. doi: 10.1093/ejo/cji122. Epub 2006 Jun 13. PMID 16772315
- [Result] Deeb R, Judge P, Peterson E, Lin JC, Yaremchuk K. Snoring and carotid artery intima-media thickness. Laryngoscope. 2014 Jun;124(6):1486-91. doi: 10.1002/lary.24527. Epub 2014 Jan 28. PMID 24242702
- [Result] Johnston CD, Gleadhill IC, Cinnamond MJ, Peden WM. Oral appliances for the management of severe snoring: a randomized controlled trial. Eur J Orthod. 2001 Apr;23(2):127-34. doi: 10.1093/ejo/23.2.127. PMID 11398550
- [Result] Ramar K, Dort LC, Katz SG, Lettieri CJ, Harrod CG, Thomas SM, Chervin RD. Clinical Practice Guideline for the Treatment of Obstructive Sleep Apnea and Snoring with Oral Appliance Therapy: An Update for 2015. J Clin Sleep Med. 2015 Jul 15;11(7):773-827. doi: 10.5664/jcsm.4858. PMID 26094920